CLINICAL TRIAL: NCT05516628
Title: Deep, Multi-omics Phenotyping to Predict Response, Resistance and Recurrence to Adjuvant Atezolizumab Plus Bevacizumab in Resected Hepatocellular Carcinoma (HCC)
Brief Title: Deep, Multi-omics Phenotyping to Predict Response, Resistance and Recurrence to Adjuvant Atezolizumab Plus Bevacizumab in Resected Hepatocellular Carcinoma
Acronym: EMPHASIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other); National University Hospital, Singapore (Other); Changi General Hospital (Other); Sengkang General Hospital (Other); Tan Tock Seng Hospital (Other); Singapore Clinical Research Institute (Other); Genome Institute of Singapore (Other); Institute of Molecular and Cell Biology of Singapore (Unknown); Cancer Science Institute of Singapore (Unknown); Duke-NUS Graduate Medical School (Other); Singapore Phenome Centre (Unknown); Nanyang Technological University (Other); NMRC OF-LCG (OFLCG21Jun-0016) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHCC12
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma (HCC); Adjuvant Atezolizumab; Adjuvant Bevacizumab; Biomarkers; Multiomics profiles; Spatial TME profiles; Surgically resected HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery followed by Adjuvant Atezolizumab-Bevacizumab Therapy every 3-weekly (Experimental): Patient will receive adjuvant Atezolizumab plus Bevacizumab every 3-weekly for two years following surgery.
  Interventions: Procedure: Surgical Resection; Drug: Adjuvant Atezolizumab-Bevacizumab Therapy

INTERVENTIONS:
Procedure: Surgical Resection — Resection of Primary Hepatocellular Cancer Tumour.
Drug: Adjuvant Atezolizumab-Bevacizumab Therapy — Patient receives adjuvant Atezolizumab plus Bevacizumab every 3-weekly for two years following resection of hepatocellular carcinoma tumour.

SUMMARY:
Hepatocellular carcinoma (HCC) is the 7th most common cancer worldwide but is the 4th deadliest, because diagnosis tend to be late and current systemic therapies are poorly efficacious. Within the same tumour, different parts of the HCC can belong to separate molecular sub-groups. In addition, there is currently no validated predictive biomarkers to help clinicians select the best therapy for an individual patient. This challenge poses an urgent, unmet clinical need.

To address this, the multi-disciplinary research program Precision Medicine in Liver Cancer across an Asia-Pacific Network (PLANet 1.0) was conceptualized and successfully conducted from 2016-22. The program uncovered novel insights into the highly heterogeneous molecular landscape of HCC and novel mechanisms, including how HCC reverts to fetal forms to escape the body's immunological defence.

These investigations will be continued in PLANet 2.0 and in this new phase, the research team will investigate patients receiving best-in-class therapeutics in 2 investigator-initiated clinical studies (AHCC12 and AHCC13), including Atezolizumab plus Bevacizumab (Atezo+Bev) and Yttrium-90, which allows the research team to collect longitudinal, before and after treatment biosamples and clinical data. These clinical studies will serve as proof-of-concept to the study team's translational findings and allow it to uncover predictive biomarkers which will help clinicians to institute more efficacious and personalized treatment in the future. The research team comprises of experts in different complementary fields (epigenomics, genomics, immunomics, metabolomics, proteomics, clinical science and data science) and across different institutions. This allows the team to adopt an integrative approach in understanding the landscape of the HCC tumour micro-environment and biomarkers co-localisation, and their role in tumour evolution and therapeutic response. By adopting a wide spectrum of converging investigations, PLANet 2.0 will identify and validate biomarkers that correlate with clinical outcomes (response, resistance and recurrence).

DETAILED DESCRIPTION:
This is a clinical translational study on a prospective, interventional clinical cohort (defined as the AHCC12 study). Patients at high risk of HCC recurrence will receive adjuvant Atezolizumab plus Bevacizumab every 3-weekly for two years following surgery. Serially collected biosamples will be deeply-phenotyped and correlated with treatment outcomes (recurrence vs non-recurrence).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing, able and mentally competent to provide written informed consent prior to any testing undertaken for this study protocol, including screening tests and evaluations that are not considered to be part of the patient's routine care.
2. Male and female patients, age 21 to 90 at the time of signature of the informed consent form.
3. Patient is able to comply with scheduled visits, assessments and other study procedures.
4. Patient diagnosed with HCC or its histological variants who has undergone a resection within 4-12 weeks prior to Day 1 of Cycle 1.

   * Multimodality treatment is not permitted, for example resection and ablation
   * Combination treatment is not permitted.
5. Patient has clinically AND histologically proven HCC after liver resection as described below:

   * Patients must have documented histological HCC confirmation of negative surgical margins (R0) which is documented in a pathology report (patients with microscopically positive [R1] or grossly positive [R2] resection margins or unknown margins will be excluded from the study).
   * Patients must have disease-free status documented within 4 weeks prior to Day 1 of Cycle 1 by a complete physical examination and radiographic images, with no subsequent evidence of residual or recurrent disease prior to Day 1 of Cycle 1. A complete set of baseline (post-resection) radiographic images and accompanying report must be available prior to Day 1 of Cycle 1.
6. Patient has an absence of major macrovascular (gross vascular) invasion of the portal vein (Vp3 or Vp4) or major macrovascular invasion in the inferior vena cava (Vv3).
7. Patient has an absence of extrahepatic spread as confirmed by CT or MRI scan of the chest, abdomen, pelvis, and head prior to and following resection . If head scan was not performed prior to resection, this must be performed after resection.
8. Patient has a full recovery from surgical resection within 4 weeks prior to Day 1 of Cycle 1.
9. Patient is at high risk for HCC recurrence after resection as defined below:

   * Tumour confined to the liver that is (i) beyond the 'up-to-7' criteria, as defined as the sum of the diameter of the largest tumour (in cm) and the number of tumours, or (ii) with macrovascualr invasion (Vp1 or Vp2).
   * In the event that the pathology and the pre- resection radiology report are discordant with regards to tumour size and number, the modality demonstrating the largest tumour size and number should be used to determine high risk features. If macrovascular invasion of Vp1 or Vp2 is detected on either the pre-operative CT/MRI scan or the pathology report, this should be a high-risk feature
10. Patient is known to be negative for the Human Immunodeficiency Virus (HIV).
11. Patient with documented virology status of hepatitis, as confirmed by screening HBV and HCV tests

    * For patients with active HBV: HBV DNA < 500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to Day 1 of Cycle 1 and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir). Patients with HBV DNA > 500 IU/mL should be continued on antiviral treatment to obtain HBV DNA < 500 IU/mL before Day 1 of Cycle 1. Antiviral treatment shall continue throughout the entire Atezo+Bev treatment phase.
    * Patients with HCV, either with resolved infection (as evidenced by detectable antibody) or chronic infection (as evidenced by detectable HCV RNA), are eligible
    * For patients with detectable HCV RNA and for whom HCV treatment is deemed appropriate by the investigator, treatment should begin no sooner than 6 months following resection consistent with AASLD guidelines
12. Patient is willing to receive an esophagogastroduodenoscopy, either before resection as part of pre-procedure work-up or following resection, and assessment and treatment of varices of all sizes per local standard of care prior to Day 1 of Cycle 1.
13. Patient is willing to receive an electrocardiogram, either before resection as part of pre-procedure work-up or following resection, prior to Day 1 of Cycle 1.
14. Patient with Child-Pugh A (up to 6 points) without clinical ascites before surgery
15. Patient with ECOG performance status 0-1.
16. Patient has adequate hematological, renal and hepatic function, defined by the following laboratory test results, obtained within 7 days prior to Day 1 of Cycle 1 unless otherwise specified:

    * AST, ALT, and ALP ≤ 5 × ULN
    * Serum bilirubin ≤ 3 × ULN
    * Albumin ≥ 28 g/L (2.8 g/dL)
    * Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 30 mL/min (calculated using the Cockcroft-Gault formula)
    * Hemoglobin ≥ 90 g/L (9 g/dL) Patients may be transfused to meet this criterion.
    * Platelet count ≥ 75 × 10**9/L (75,000/µL) without transfusion
    * Lymphocyte count ≥ 0.5 × 10**9/L (500/µL)
    * ANC ≥ 1.5 × 10**9/L (1500/µL) without granulocyte colony-stimulating factor support
    * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 2 × ULN
    * Urine dipstick for proteinuria < 2 + (within 7 days prior to Day 1 of Cycle 1) Patients discovered to have ≥ 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection (or an alternative method such as protein:creatinine ratio, per local guidance) and must demonstrate < 1 g of protein in 24 hours.
17. Patient is estimated to have a life expectancy of at least 3 months without any active treatment.
18. Patient is deemed suitable for protocol treatment as determined by clinical assessment undertaken by the site Investigator.
19. (For female patients) Patient is either postmenopausal or, if premenopausal, must have a negative pregnancy test and agree to use two forms of contraception if sexually active during the treatment period, for at least 5 months after the last dose of atezolizumab and 6 months after the last dose of bevacizumab.
20. (For male patients) Patient is surgically sterile, or if sexually active and having a pre-menopausal female partner, must be using an acceptable form of contraception during the treatment period and for 6 months after the last dose of bevacizumab.

Exclusion Criteria:

1. Patient is unable to provide informed consent or refuse blood taking.
2. Patient has evidence of residual, recurrent, or metastatic disease prior to initiation of treatment.
3. Patient has clinically significant ascites or any other clinical signs of liver failure on physical examination at time of enrolment.
4. Patient has a history of hepatic encephalopathy.
5. Patient has a bleeding event due to untreated or incompletely treated esophageal and/or gastric varices prior to Day 1 of Cycle 1.
6. Patient has active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     * Rash must cover < 10% of body surface area.
     * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
     * There is no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the 12 months prior to Day 1 of Cycle 1.
7. Patient has a history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on chest CT scan at screening.
8. Patient has significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to Day 1 of Cycle 1, unstable arrhythmia, or unstable angina
9. Patient has a history of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer. Effectively treated malignancies,including HCC that have been in remission for over 5 years can be allowed as they are highly likely to have been cured.
10. Patient has active tuberculosis at screening
11. Patient has a severe infection within 4 weeks prior to Day 1 of Cycle 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that in the opinion of the investigator, could impact patient safety
12. Patient has received treatment with therapeutic oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1

    • Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
13. Patient has prior allogeneic stem cell or solid organ transplantation
14. Patient is on the waiting list for liver transplantation
15. Patient has any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
16. Patient has a co-infection with HBV and HCV or Hepatitis D viral infection

    • Patients with a history of HCV infection but who are negative for HCV RNA by polymerase chain reaction will be considered to be negative for HCV infection.
17. Patient has clinically significant uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12mg/dL, or corrected serum calcium > ULN)
18. Patient has a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
19. Patient has known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulations
20. Patient has received any treatment for HCC prior to resection, including previous liver resection, systemic therapy (including investigational agents) and locoregional therapy (e.g. RFA, TACE, SIRT), radiotherapy, immunotherapy, chemotherapy or neo-adjuvant chemotherapy other than the planned surgery. However, patient who has received previous HCC resection more than 5 years ago is deemed to have a de-novo liver tumour and therefore can be included.

    * Prior use of herbal therapies or traditional Chinese medicines with anti-cancer activity included in the label is allowed, but such therapies must be discontinued at least 7 days prior to Day 1 of Cycle 1 and are prohibited during the study.
    * Portal vein embolization used to increase the functional liver remnant prior to surgery is permitted.
21. Patient has received or plans to receive treatment with a live, attenuated vaccine within 4 weeks prior to Day 1 of Cycle 1, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
22. Patient has received prior treatment with investigational therapy within 4 weeks prior to Day 1 of Cycle 1
23. Patient has prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
24. Patient has received prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to Day 1 of Cycle 1
25. Patient has received prior treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor-α [TNF-α] agents) within 2 weeks prior to Day 1 of Cycle 1, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
26. Patient has inadequately controlled arterial hypertension (defined as systolic blood pressure [BP] > 150 mmHg and/or diastolic BP > 100 mmHg), based on an average of at least three BP readings at two or more sessions

    • Anti-hypertensive therapy to achieve these parameters is allowed.
27. Patient has a history of hypertensive crisis or hypertensive encephalopathy
28. Patient has significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of Cycle 1
29. Patient has a history of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to Day 1 of Cycle 1
30. Patient has evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
31. Current or recent (within 10 days prior to Day 1 of Cycle 1) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose

    * Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 × ULN and aPTT is within normal limits (according to institutional standards) within 14 days prior to Day 1 of Cycle 1.
    * Prophylactic use of low-molecular-weight heparin (LWMH; i.e., enoxaparin 40 mg/day) is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk. Benefits and risks should be assessed and caution exercised for use of direct oral anticoagulants. The investigator should consider switching to other approved anticoagulants due to the risk of upper GI bleeding in patients with HCC.
32. Patient has received a core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to Day 1 of Cycle 1
33. Patient has a history of GI fistula, GI perforation, or intra-abdominal abscess within 6 months prior to Day 1 of Cycle 1
34. Patient has evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
35. Patient has a serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
36. Patient is receiving or plans to receive a major surgical procedure within 4 weeks prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure during the study
37. Patient has a history of clinically significant intra-abdominal inflammatory process within 6 months prior to Day 1 of Cycle 1, including, but not limited to, peptic ulcer disease, diverticulitis, or colitis
38. (For female patients) Patient is pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of atezolizumab or within 6 months after the final dose of bevacizumab

    * Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to Day 1 of Cycle 1.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free-survival (RFS) in relation to the multi-omics (epigenomics, genomics, transcriptomics, proteomics and metabolomics) and spatial TME profiles of both tissue and peripheral blood. | Up to 4 Years after surgery.
  Biomarkers that are predictive of response to study treatment based on the multi-omics (epigenomics, genomics, transcriptomics, immunomics, proteomics and metabolomics) and spatial TME profiles of both tissue and peripheral blood.

SECONDARY OUTCOMES:
Proportion of patients who are amenable to surgical resection upon recurrence following adjuvant therapy. | Up to 4 Years after surgery.
Time to Recurrence (TTR) after surgery. | Up to 4 Years after surgery.
  The time from date of surgery to the first documented occurrence of intrahepatic or extrahepatic HCC.
Time to Recurrence (TTR) after treatment. | Up to 4 Years after surgery.
  The time from start date of treatment to the first documented occurrence of intrahepatic or extrahepatic HCC.
Recurrence Free Survival (RFS) after surgery. | Up to 4 Years after surgery.
  The time from date of surgery to the first documented occurrence of intrahepatic or extrahepatic HCC, or death (whichever occurs first).
Recurrence Free Survival (RFS) after treatment. | Up to 4 Years after surgery.
  The time from start date of treatment to the first documented occurrence of intrahepatic or extrahepatic HCC, or death (whichever occurs first).
Overall Survival (OS). | Up to 4 Years after surgery.
  The time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce CHOW, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (6):
- Singapore (6):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No